CLINICAL TRIAL: NCT06595602
Title: Intelligent Lung Support in the Intensive Care Unit (IntelliLung): An Observational, Prospective, Multicentre Study
Brief Title: Intelligent Lung Support in the Intensive Care Unit
Acronym: IntelliLung
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: Dipartimento di Scienze Chirurgiche e Diagnostiche Integrate, University of Genoa, Genoa, Italy (Unknown); Critical Care Department, Parc Taulí Hospital Universitari, Institut d'Investigació I Innovació Parc Taulí (I3PT-CERCA), Sabadell, Spain (Unknown); Department of Anaesthesiology and Intensive Care, National Medical Institute of the Ministry of Interior and Administration, Warsaw, Polan (Unknown); Department of Intensive Care Medicine. Hospital Universitario de La Princesa. Universidad Autonoma de Madrid, Madrid, Spain (Unknown); Department of Anesthesiology and Intensive Care Medicine, Pulmonary Engineering Group, Faculty of Medicine and University Hospital Carl Gustav Carus, TUD Dresde (Unknown)
Responsible Party: Sponsor
Other Study IDs: TUD-INTELL-086; 101057434 (Other Grant/Funding Number: European Union)
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Mechanical Ventilation; Intensive Care Medicine
Keywords: Invasive mechanical ventilation; Intensive care medicine; critical care medicine; artificial intelligence; decision support

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Invasively mechanically ventilated patients expected to stay ventilated for more than 24 h.
  Interventions: Device: Artificial intelligence based decision support system (AI-DSS); software

INTERVENTIONS:
Device: Artificial intelligence based decision support system (AI-DSS); software — The device is intended for monitoring and recommending ventilator settings, ventilation mode to qualified Intensive Care Unit (ICU) health care professionals (HCP). This is for medical indications that require invasive mechanical ventilation of the respiratory system in the ICU under international / EU guidelines.
  The device receives clinical data via the ICU's data integration platform that includes patient physical and demographic data as well as current vital signs, ventilation parameters, blood gas analysis, general blood laboratory reports, fluid balance and medication. Prediction models based on artificial intelligence algorithms are used to deduce therapy suggestions from received data. The algorithm is carried out on a secured cloud platform.

SUMMARY:
The aim of this observational study is to test the IntelliLung decision support system based on artificial intelligence. This system is intended to help to set the ventilator. The study includes patients with and without ARDS (acute respiratory distress syndrome) who are receiving invasive mechanical ventilation, as well as patients with additional extracorporeal lung support. The study will be conducted in several centers.

The main question of the study:

How well do the mechanical ventilation settings of healthcare staff match the recommendations of the IntelliLung system?

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients, age ⪰18 years
2. Written informed consent
3. Invasively mechanically ventilated patients expected to be intubated for more than 24 hours.

Exclusion Criteria:

1. Expected to die within ≤48 hours
2. Participation in an interventional mechanical ventilation trial
3. Mechanical Ventilation with a closed-loop ventilation mode
4. Persons dependent on the sponsor and/or investigator
5. Subjects who are currently imprisoned or otherwise in confinement ordered by law or other official authorities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Invasively mechanically ventilated, adult, acute respiratory distress syndrome (ARDS) and non-ARDS patients expected to stay intubated and ventilated for more than 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 530 (Estimated)
Dates: Start 2025-05-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Relative time of same device settings of healthcare provider and IntelliLung AI-DSS related to the total IntelliLung AI-DSS running time | From enrollment to discharge from the intensive care unit or successful weaning from the ventilator, assessed up to 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Wittenstein, Principal Investigator — epartment of Anesthesiology and Intensive Care Medicine, Pulmonary Engineering Group, Faculty of Medicine and University Hospital Carl Gustav Carus, TUD Dresden University of Technology, Dresden, Germany
Locations (5):
- Department of Anesthesiology and Intensive Care Medicine, Pulmonary Engineering Group, Faculty of Medicine and University Hospital Carl Gustav Carus, TUD Dresden University of Technology, Dresden, Germany, Dresden, Germany
- Dipartimento di Scienze Chirurgiche e Diagnostiche Integrate, University of Genoa, Genoa, Italy, Genova, Italy
- Department of Anaesthesiology and Intensive Care, National Medical Institute of the Ministry of Interior and Administration, Warsaw, Poland, Warsaw, Poland
- Spain (2):
  - Department of Intensive Care Medicine. Hospital Universitario de La Princesa. Universidad Autonoma de Madrid, Madrid, Spain, Madrid
  - Critical Care Department, Parc Taulí Hospital Universitari, Institut d'Investigació I Innovació Parc Taulí (I3PT-CERCA), Sabadell, Spain, Sabadell

IPD SHARING:
Plan to Share IPD: Undecided